CLINICAL TRIAL: NCT02168491
Title: Feasibility of Once-daily Administered GLP-1 Receptoragonist (Lixisenatide) in Combination With Basal Insulin in Patients With Type-2 Diabetes Mellitus Not Achieving Therapeutic Targets With Premixed Insulin
Brief Title: Feasibility of Once/Daily Administered GLP/1 Receptoragonist (Lixisenatide) in Combination With Basal Insulin
Acronym: LixiBIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Prof. MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LixiBIT_V3; 2013-005334-37 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental): 10 type 2 diabetic patients will be included to perform in this study and will be switched from premixed insulin to insulin glargine and lixisenatide
  Interventions: Drug: Lixisenatide; Drug: Insulin glargine

INTERVENTIONS:
Drug: Lixisenatide — Patients will be switched to basal insulin glargine (Lantus, once daily in the morning) and GLP-1 receptor agonist Lixisenatide (Lyxumia, once daily in the morning before breakfast; days 1-14 10 µg thereafter 20 µg). The (mean) daily dose of premixed insulin will be calculated based on the records of the run in period. The initial dose of insulin glargine will be adjusted at about 60% of the daily insulin dose of premixed insulin. This is based on the observed reduction of required insulin dose described in recent literature upon initiation with a GLP-1 agonist.
  Other Names: Lyxumia
Drug: Insulin glargine — Patients will be switched to basal insulin glargine (Lantus, once daily in the morning) and GLP-1 receptor agonist Lixisenatide (Lyxumia, once daily in the morning before breakfast; days 1-14 10 µg thereafter 20 µg). The (mean) daily dose of premixed insulin will be calculated based on the records of the run in period. The initial dose of insulin glargine will be adjusted at about 60% of the daily insulin dose of premixed insulin. This is based on the observed reduction of required insulin dose described in recent literature upon initiation with a GLP-1 agonist.
  Other Names: Lantus

SUMMARY:
Premixed insulin-based therapy is a standard insulin treatment strategy in Austria. The widespread use of premixed insulin is explained by high acceptance by health care professionals and patients due to one single product and flexible number of injections (1-3 daily) which covers the demand in controlling fasting and postprandial glucose excursions of most patients with diabetes. However, the use of pre-mixed insulin frequently leads to a high insulin demand and consequently weight gain and an increased risk of hypoglycemia. Hence, achieve good metabolic control in these patients remains a major challenge.

For those patients, the approach to treatment intensification without facing the typical risks of insulin treatment (hypoglycemia and weight increase) is of major importance. One, so far not exploited option may be the BIT-strategy: Basal insulin in combination with incretin-based therapy.

Pathophysiologically basal insulin inhibits glucose production in the liver, decreases hepatic insulin resistance and improves the function of beta cells in the postprandial state by discharge of fasting insulin secretion. During further diabetes progression steadily increasing HbA1c levels - despite good fasting blood glucose control - indicate the need for additional intervention of meal-related glucose excursions. In this stage of type-2 diabetes basal insulin can be combined with prandial (short-acting) insulin or prandial GLP-1 receptor agonists. However, regarding important safety parameters: risks of hypoglycemia and weight gain in the long-term treatment GLP-1 receptor agonists are beneficial.

Lixisenatide is a novel GLP-1 receptor agonist with a pronounced postprandial (PPG) effect which fits with basal insulin mode of action primarily focused on fasting blood glucose reduction.

Therefore 10 patients (both gender) under treatment with premixed insulin (2-3 times daily) and HbA1c>7% will be switched to basal insulin glargine (Lantus, once daily) and GLP-1 receptor agonist Lixisenatide (Lyxumia, once daily). The investigators hypothesize that switching from a therapy based on premixed insulin to a simple, once daily administered combination of basal insulin plus a GLP-1 receptor agonist in patients with type-2 diabetes not achieving therapeutic target (HbA1c>7%) is clinically feasable in an out patient setting

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70a
* Subjects understand study related activities and give written informed concent
* HbA1c between 7 - 10 % under treatment with premixed insulin (2-3 injections)

Exclusion Criteria:

* Females of child-bearing age
* History of hypoglycemia unawareness
* Gastrointestinal disease associated with prolonged nausea and vomiting
* Impaired liver function (transaminase >2x than normal)
* Impaired kidney function (creatinin > 1,2 mg/dl)
* Known intolerance against GLP-1 receptor agonists
* History of pancreatitis or pancreas tumor
* Malignancies, autoimmune diseases
* Severe dyslipidemia (serum triglycerides > 400 mg/dl, cholesterol > 300 mg/dl)
* Psychiatric disorder
* Oral glucose lowering medication except for metformin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krebs, MD, Prof., Principal Investigator — Medical University of Vienna, Währinger Gürtel 18-20, 1090 Vienna, Austria
Locations (1):
- Medical University Of Vienna, Department of Internal Medicine III, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Harreiter J, Kosi-Trebotic L, Lukas A, Wolf P, Winhofer Y, Luger A, Kautzky-Willer A, Krebs MR. Switch to Combined GLP1 Receptor Agonist Lixisenatide with Basal Insulin Glargine in Poorly Controlled T2DM Patients with Premixed Insulin Therapy: A Clinical Observation and Pilot Study in Nine Patients. Diabetes Ther. 2017 Jun;8(3):683-692. doi: 10.1007/s13300-017-0249-4. Epub 2017 Mar 29. PMID 28357772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were screened
Pre-assignment Details: 2 patients declined to participate because of time restraints, thus study medication was administered in 9 patients
Groups:
- Lixisenatide With Basal Insulin (LixiBIT): Type 2 diabetic patients will be included to perform in this study and will be switched from premixed insulin to insulin glargine and lixisenatide
  Lixisenatide: Patients will be switched to basal insulin glargine (Lantus, once daily in the morning) and GLP-1 receptor agonist Lixisenatide (Lyxumia, once daily in the morning before breakfast; days 1-14 10 µg thereafter 20 µg). The (mean) daily dose of premixed insulin will be calculated based on the records of the run in period. The initial dose of insulin glargine will be adjusted at about 60% of the daily insulin dose of premixed insulin. This is based on the observed reduction of required insulin dose described in recent literature upon initiation with a GLP-1 agonist.
  Insulin glargine: Patients will be switched to basal insulin glargine (Lantus, once daily in the morning) and GLP-1 receptor agonist Lixisenatide (Lyxumia, once daily in the morning before breakfast; days 1-14 10 µg thereafter 20 µg). The (mean) daily dose of
Period: Overall Study
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Lixisenatide With Basal Insulin (LixiBIT): Type 2 diabetic patients will be included to perform in this study and will be switched from premixed insulin to insulin glargine and lixisenatide
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to End
Description: A change between two time points is reported. Time Frame: baseline and 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: HbA1c in percent
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Number analyzed (Participants) | 9
HbA1c in percent | -0.54 (0.52)
Statistical Analysis 1: Comparison: Lixisenatide With Basal Insulin (LixiBIT); Test type: Superiority or Other; p < 0.02, paired t test

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG, Mean Over 2 Weeks)
Description: Patients will be instructed to record all insulin injections and a complete 7-point-blood glucose profile (fasting, 2h after breakfast, before lunch, 2h after lunch, before dinner, 2h after dinner, late before going to bed) during a one-week prestudy run-in period to confirm compliance and document current metabolic control and doses of premixed insulin.
  Patients will be asked to record not only glucose profiles (at least 4 measurements per day) but also the occurrence of hypoglycemic symptoms or other adverse effects daily throughout the study.
  During the last week of the study patients will be asked to again record a complete 7-point-blood glucose profile (fasting, 2h after breakfast, before lunch, 2h after lunch, before dinner, 2h after dinner, late before going to bed) and drug injections to confirm compliance and document metabolic control.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: glucose in mg/dl
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Number analyzed (Participants) | 9
glucose in mg/dl | -9 [-24.1 to 6.1]
Statistical Analysis 1: Comparison: Lixisenatide With Basal Insulin (LixiBIT); Test type: Superiority or Other; p = 0.24, paired t test

3. Secondary Outcome: Change in Body Weight From Baseline to End of Study
Description: A change between two time points is reported. Time Frame: baseline and 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: weight in kg
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Number analyzed (Participants) | 9
weight in kg | -1.4 (3.6)
Statistical Analysis 1: Comparison: Lixisenatide With Basal Insulin (LixiBIT); Test type: Superiority or Other; p = 0.28, paired t test

ADVERSE EVENTS:
Arm/Group | Lixisenatide With Basal Insulin (LixiBIT)
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lixisenatide With Basal Insulin (LixiBIT) (N=9)
elective ENT surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lixisenatide With Basal Insulin (LixiBIT) (N=9)
mild asymptomatic hypoglycaemia (Endocrine disorders) | 3 (8)
mild gastrointestinal complaints (Gastrointestinal disorders) | 2 (3)
urinary tract infection (Infections and infestations) | 2 (3)
symptomatic hypoglycaemia (Endocrine disorders) | 1 (1)
hypercholesterolaemia (Endocrine disorders) | 2 (2)
haematuria (Renal and urinary disorders) | 1 (1)
cough (General disorders) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
elective ambulatory cataract surgery (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No